CLINICAL TRIAL: NCT04269707
Title: Evaluating the Efficacy and Safety of Intravenous Ferric Carboxymaltose in Pediatric Patients With Iron Deficiency Anemia and an Unsatisfactory Response to Oral Iron Under Study Protocol 1VIT17044
Brief Title: Efficacy and Safety of Intravenous Ferric Carboxymaltose in Pediatric Patients With Iron Deficiency Anemia and Unsatisfactory Response Oral Iron Under Study Protocol 1VIT17044
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT18045
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Results first posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: This is a single arm, open-label, multi-center, multi-national, non-randomized study that will evaluate the efficacy and safety of a one course treatment with FCM in participants who had an unsatisfactory response to oral iron in study 1VIT17044.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IV Iron (Other): The primary objective in this study is to allow participants who were randomized to receive oral iron in the 1VIT17044 trial and who had an unsatisfactory response to oral iron or those that required a concomitant intervention, (defined as, blood transfusion, use of IV or oral iron outside of protocol, increase in erythropoietin for any reason [Day 0 thru Day 35 of study protocol 1VIT17044], change in IBD treatment) to receive one course of FCM. This course of FCM will consist of two doses of FCM at 15 mg/kg (maximum single dose of 750 mg), separated by seven days.
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Ferric carboxymaltose — IV iron

SUMMARY:
Evaluating the Efficacy and Safety of Intravenous Ferric Carboxymaltose in Pediatric Patients with Iron Deficiency Anemia and an Unsatisfactory Response to Oral Iron under Study Protocol 1VIT17044

DETAILED DESCRIPTION:
This is a single arm, open-label, multi-center, multi-national, non-randomized study that will evaluate the efficacy and safety of a one course treatment with FCM in participants who had an unsatisfactory response to oral iron in study 1VIT17044.

Subjects will have an End of Study (EOS) Visit (Day 35) from the 1VIT17044 study to qualify for entry. Subjects will then be screened, meet all inclusion criteria, no exclusion criteria and have a baseline evaluation. Based on the successful completion of the baseline evaluations, subjects will be enrolled and will receive the first dose of FCM (Day 0). The second FCM dose will occur 7 days from the first dose. Subjects will return to the clinic 14 and 28 days post their first dose for laboratory and safety assessments, and at 35 days post the first dose, participants will return to the clinic for final safety and efficacy assessments. Once all assessments are complete the participant will exit the study.

An unsatisfactory response to oral iron (i.e., an increase in hemoglobin (Hgb) of <1 g/dL from baseline) will be defined as non-responders to oral iron treatment. Non-responders who continue to meet all inclusion criteria (including Hgb <11 g/dL) and none of the exclusion criteria will receive 1 course of FCM.

ELIGIBILITY:
Inclusion Criteria:

1. Unsatisfactory response to oral iron or those that required a concomitant intervention, (defined as, blood transfusion, use of IV or oral iron outside of protocol, increase in erythropoietin for any reason [Day 0 thru Day 35 of study protocol 1VIT17044], change in IBD treatment).
2. Hgb <11 g/dL
3. Ferritin ≤300 ng/mL and TSAT <30%

Exclusion Criteria:

1. Known history of hypersensitivity reaction to any component of FCM.
2. History of acquired iron overload, hemochromatosis, or other iron accumulation disorders.
3. History of significant diseases of the liver, hematopoietic system, cardiovascular system, psychiatric disorder, or other conditions which, in the opinion of the investigator, may place a subject at added risk for participation in the study.
4. Any existing non-viral infection.
5. Known history of positive HBsAg or HCV with evidence of active hepatitis.
6. Known history of positive HIV-1/HIV-2 antibodies (anti-HIV).
7. Anemia due to reasons other than iron deficiency (e.g., hemoglobinopathy and vitamin B12 or folic acid deficiency) that has not been corrected.
8. Administration and / or use of an investigational product (drug or device) within 30 days of screening.
9. Alcohol or drug abuse within the past six months.
10. Female participant who is pregnant or lactating, or sexually active females who are of childbearing potential not willing to use an acceptable form of contraceptive precautions during the study.
11. Unable to comply with study procedures and assessments.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Falone, MD, Study Director — American Regent, Inc.
Locations (2):
- United States (2):
  - Miami Clinical Research, Miami, Florida
  - South Florida Research Phase I-IV, Miami Springs, Florida

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1VIT17044, NCT03523117 can be referenced to make the information accessible.
Groups:
- IV Iron: The primary objective in this study is to allow participants who were randomized to receive oral iron in the 1VIT17044 trial and who had an unsatisfactory response to oral iron or those that required a concomitant intervention, (defined as, blood transfusion, use of IV or oral iron outside of protocol, increase in erythropoietin for any reason [Day 0 thru Day 35 of study protocol 1VIT17044, NCT03523117 can be referenced to make the information accessible.], change in IBD treatment) to receive one course of FCM. This course of FCM will consist of two doses of FCM at 15 mg/kg (maximum single dose of 750 mg), separated by seven days.
  Ferric carboxymaltose: IV iron
Period: Overall Study
Arm/Group | IV Iron
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IV Iron
Number analyzed (Participants) | 7
Age, Customized [Count of Participants; unit: Participants]
  Age | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin From Baseline to Day 35
Description: The change in hemoglobin from Baseline to Day 35 was assessed using paired t-tests (two-sided test, α = 0.05). Baseline hemoglobin was defined as the last hemoglobin obtained before the first dose.
Time Frame: The change in Hgb from baseline to day 35
Population: The change in hemoglobin from Baseline to Day 35 was assessed using paired t-tests (two-sided test, α = 0.05). Baseline hemoglobin was defined as the last hemoglobin obtained before the first dose.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | IV Iron
Number analyzed (Participants) | 7
g/dL | 0.70 [-0.40 to 1.80]
Statistical Analysis 1: Comparison: IV Iron; Test type: Non-Inferiority — Change in hemoglobin from baseline to day 35 was assessed using paired t-tests (two-sided test, alpha = 0.05); p = 0.1711, t-test, 2 sided; Mean Difference (Final Values) = 0.70, 95% CI 2-sided [-0.40 to 1.80]

ADVERSE EVENTS:
Time Frame: Day 1 through Day 35
Description: AE will be elicited by nonspecific questions such as "Have you noticed any problems?" Participants will be encouraged to report adverse events at their onset.
  Any AE spontaneously reported by, elicited from the participant, or observed by the physician or study staff, shall be recorded on the appropriate AE page of the eCRF. The investigator will record the date and time of onset, severity, the relationship to study medication, the date and time of resolution and the outcome of the AE.
Arm/Group | IV Iron
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT04269707/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT04269707/SAP_001.pdf